CLINICAL TRIAL: NCT01816321
Title: Corifollitropin Alfa Followed by Hp-HMG Versus Recombinant FSH in Young Poor Ovarian Responders. A Multicentre Randomized Controlled Clinical Trial
Brief Title: Corifollitropin Alfa Followed by Menotropin for Poor Ovarian Responders Trial
Acronym: COMPORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nikolaos P. Polyzos, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 143201316398; 2013-000583-29 (EudraCT Number)
Record Dates: First submitted 2013-03-16; First posted 2013-03-22 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Infertility; Poor Ovarian Response
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corifollitropin alfa followed by hpHMG (Experimental)
  Interventions: Drug: Corifollitropin alfa; Drug: Ganirelix; Drug: hp HMG
- recombinant FSH (Active Comparator)
  Interventions: Drug: recombinant FSH; Drug: Ganirelix

INTERVENTIONS:
Drug: Corifollitropin alfa — Corifollitropin alfa 150μg on day 2 of the menstrual cycle (stimulation day 1)
  Arms: Corifollitropin alfa followed by hpHMG
Drug: recombinant FSH — recombinant FSH 300IU/daily from day 2 of the cycle (stimulation day 8)until day of ovulation triggering
  Arms: recombinant FSH
Drug: Ganirelix — Ganirelix 0.25mg/daily from day 7 of the cycle(stimulation day 6) until day of ovulation triggering
Drug: hp HMG — hp HMG 300IU/daily from day 9 of the cycle (stimulation day 8)until day of ovulation triggering
  Arms: Corifollitropin alfa followed by hpHMG

SUMMARY:
In combination with the existing literature, previous work indicates that 1) women with poor ovarian response fulfilling the "Bologna criteria" have very low pregnancy rates, irrespective of age 2) current treatment protocols demonstrate ongoing pregnancy rates that do not exceed 8.5% and 3) corifollitropin alfa followed by hpHMG might increase ongoing pregnancy rates in young patients (<40years old) fulfilling the criteria. These findings provide a strong rationale for a definitive large RCT. The COMPORT study will provide conclusive evidence regarding the superiority or not of this novel protocol with corifollitropin alfa followed by hpHMG for the treatment of young poor ovarian responders fulfilling the Bologna criteria.

DETAILED DESCRIPTION:
Recently, the European Society of Human Reproduction and Embryology developed a new definition in order to select patients suitable for inclusion in future clinical trials as poor ovarian responders, the so-called "Bologna criteria". However, a limited number of studies has been published to date including patients with poor ovarian response according to the "Bologna criteria", whereas no randomized trial is published or ongoing for this population.

Preliminary reports in "Bologna poor responders" highlight the limited prospects for these women. Natural cycle IVF has been shown to result in disappointingly low live birth rates, regardless of patients' age and ovarian stimulation with widely accepted treatment modalities, e.g. short agonist protocol, did not appear demonstrate substantial benefits.

Nonetheless, despite the disappointing results from the vast majority of the preliminary studies in this population, a recent pilot study by our group has shown that a specific protocol may indeed be a promising option for women of younger age fulfilling the "Bologna criteria". Corifollitropin alfa followed by highly purified hMG in an antagonist protocol demonstrated an ongoing pregnancy rate of 28% in women <40years, strongly suggesting the conduction of a future randomized trial testing this novel treatment protocol

ELIGIBILITY:
Inclusion Criteria:

* Age less than 40 years
* Fulfillment of the "Bologna criteria" for poor ovarian response.

Based on inclusion criteria two patients' categories are eligible:

1. Women < 40 years old AND ≤3 oocytes in one of the previous cycles AND (Antral follicle count <7 or antimullerian hormone serum values <1.1 ng/ml)
2. Women <40 years old and ≤3 oocytes in two the previous cycles with maximum ovarian stimulation

In addition women less than 40 years old will be considered eligible if they had undergone previous ovarian surgery or chemotherapy (risk factors for poor ovarian response) and have an AMH<1.1ng/ml or an AFC<7, as suggested by the Bologna criteria

Exclusion Criteria:

* Uterine abnormalities
* Recent history of any current untreated endocrine abnormality
* Unilateral or bilateral hydrosalpinx (visible on transvaginal ultrasound, unless clipped)
* Contraindications for the use of gonadotropins
* Recent history of severe disease requiring regular treatment

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 9-10 weeks of gestation
  The presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity at 9-10 weeks of gestation.

SECONDARY OUTCOMES:
Clinical pregnancy | 7 weeks of gestation
  The presence of intrauterine gestational sac at 7 weeks of gestation
Biochemical pregnancy | 2 weeks after embryo transfer
  Positive pregnancy test 2 weeks after embryo transfer
Number of oocytes retrieved | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval

OTHER OUTCOMES:
Cycle cancellation due to poor ovarian response | Day 8-10 of ovarian stimulation
  Number of cycles cancelled due to monofollicular or no follicular development
Number of cycles reaching the stage of embryo transfer | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated 3 days after oocyte retrieval
Number and quality of embryos | Day of embryo transfer
  3 days after oocyte retrieval
Number of cycles with frozen supernumerary embryos | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated 5 days after oocyte retrieval or 2-3 days after embryo transfer in case of an embryo transfer
Endocrine parameters (LH,FSH, E2, Progesterone) during ovarian stimulation | Days 1,6,8,10 of stimulation and day of ovulation triggering
Cycle cancellation due to serious adverse effects of medication | 20-25 days after initiation of stimulation
  20-25 days after the initiation of ovarian stimulation all patients (cycles) will be monitored for the occurence of any adverse effect and cycle cancellation(during ovarian stimulation) due to a serious adverse effect from medication

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Polyzos NP, De Vos M, Corona R, Vloeberghs V, Ortega-Hrepich C, Stoop D, Tournaye H. Addition of highly purified HMG after corifollitropin alfa in antagonist-treated poor ovarian responders: a pilot study. Hum Reprod. 2013 May;28(5):1254-60. doi: 10.1093/humrep/det045. Epub 2013 Feb 26. PMID 23442756
- [Background] Polyzos NP, Devos M, Humaidan P, Stoop D, Ortega-Hrepich C, Devroey P, Tournaye H. Corifollitropin alfa followed by rFSH in a GnRH antagonist protocol for poor ovarian responder patients: an observational pilot study. Fertil Steril. 2013 Feb;99(2):422-6. doi: 10.1016/j.fertnstert.2012.09.043. Epub 2012 Oct 16. PMID 23084565
- [Background] Polyzos NP, Blockeel C, Verpoest W, De Vos M, Stoop D, Vloeberghs V, Camus M, Devroey P, Tournaye H. Live birth rates following natural cycle IVF in women with poor ovarian response according to the Bologna criteria. Hum Reprod. 2012 Dec;27(12):3481-6. doi: 10.1093/humrep/des318. Epub 2012 Aug 30. PMID 22940767
- [Background] Polyzos NP, Devroey P. A systematic review of randomized trials for the treatment of poor ovarian responders: is there any light at the end of the tunnel? Fertil Steril. 2011 Nov;96(5):1058-61.e7. doi: 10.1016/j.fertnstert.2011.09.048. PMID 22036048
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Derived] Drakopoulos P, Vuong TNL, Ho NAV, Vaiarelli A, Ho MT, Blockeel C, Camus M, Lam AT, van de Vijver A, Humaidan P, Tournaye H, Polyzos NP. Corifollitropin alfa followed by highly purified HMG versus recombinant FSH in young poor ovarian responders: a multicentre randomized controlled clinical trial. Hum Reprod. 2017 Nov 1;32(11):2225-2233. doi: 10.1093/humrep/dex296. PMID 29040589